CLINICAL TRIAL: NCT06067724
Title: Effect of Pelvic and Trunk Control Exercises on Function Outcome of Affected Upper Extremity in Stroke Patients
Brief Title: Effect of Pelvic Control Exercises in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rowida Abd Elgleel Sayed Abd Elgleel, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pelvic control in stroke
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic and trunk control exercises (Active Comparator): Twenty Egyptian male stroke patients will receive 40 minutes of pelvic and trunk control exercises for six weeks after a 30 minutes of traditional physical therapy program.
  Interventions: Other: Pelvic and trunk control exercises
- Traditional physical therapy (Sham Comparator): Twenty Egyptian male stroke patients will receive 30 minutes of sham traditional physical therapy program for six weeks.
  Interventions: Other: Pelvic and trunk control exercises

INTERVENTIONS:
Other: Pelvic and trunk control exercises — Patients in this group will be treated by the traditional physical therapy program in addition to a 18 sessions of pelvic and trunk control exercises for 40 min included abdominal drawing in maneuver for contraction of transversus abdominis pelvic tilting exercises and pelvic stabilization exercises from different positions. Pelvic tilting exercises included; anterior, posterior, lateral pelvic tilting and pelvic rotation on a therapeutic ball. Pelvic stabilization exercises include bridging, half bridging, clamshell from supine and side lying, quadribed exercises, weight shifting on the affected limb from standing by forward and diagonal reach out, ball bridging and rhythmic stabilization exercises

SUMMARY:
The purpose of the study is to investigate the combined effect of pelvic and trunk control exercises on muscle performance of affected upper extremity in stroke patients.

DETAILED DESCRIPTION:
The study conducted on forty stroke patients. They assessed by Biodex System 3 Pro Isokinetic, Modified Ashworth Scale(MAS), Fugel Meyer Assessment scale (FMAS), Box and block test and hand grip dynamometer. Patients divided into control group and study group. The control group treated by a traditional physical therapy program.The study group treated by the traditional physical therap program in addition to pelvic and trunk control exercises for 40 min.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age will range from 45 - 60 years.
* Muscle tone grade will range from 1 to 1+ according to modified Ashworth scale.
* Duration of illness will range from 6 to 18 months after stroke onset.
* Ability of the patient to stand without assistive devices.

Exclusion Criteria:

* • Other neurological or musculoskeletal disorders that might affect pelvic alignment such as severe arthritis, knee surgery, total hip joint replacement, lower limb fractures, contractures of fixed deformity or leg length discrepancy.

  * Severe chronic back and/or knee pain that might affected standing posture.
  * Recurrent stroke
  * Shoulder or upper limb injury that might affect the recovery.
  * Perceptual or cognitive dysfunctions.
  * BMI > 30

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-07 (Estimated)

PRIMARY OUTCOMES:
Biodex System 3 Pro Isokinetic | Six weeks after the beginning of the intervention
  Changes in peak muscle torque of upper limb muscles from baseline to four weeks after the beginning of intervention

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity | Six weeks after the beginning of the intervention
  Changes in upper limb function from baseline to four weeks after the beginning of intervention
Box and block test | Six weeks after the beginning of the intervention
  Changes in gross hand function from baseline to four weeks after the beginning of intervention
Hand grip dynamometer | Six weeks after the beginning of the intervention
  . Changes in hand grip strength from baseline to four weeks after the beginning of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy labs at Cairo University, Giza, Egypt